CLINICAL TRIAL: NCT03049098
Title: Visual Perception Exploration Using Eye-tracking Technology in High-fidelity Medical Simulation
Status: Completed | Type: Observational
Sponsor: Issam Tanoubi (Other)
Responsible Party: Sponsor-Investigator, Issam Tanoubi, Université de Montréal, Université de Montréal
Organization: Université de Montréal (Other)
Other Study IDs: MMT-2016
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Simulation Training; Perception; Eye Movements; Task Performance and Analysis
Keywords: Eye-tracking; High Fidelity Simulation Training; Visual Perception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Success at the simulation: Participant could correctly set the pacing unit to obtain electrical and mechanical pacing of the mannequin in nine minutes.
  Interventions: Behavioral: Simulation
- Failed the simulation: Participant could not correctly set the pacing unit to obtain electrical and mechanical pacing of the mannequin in nine minutes.
  Interventions: Behavioral: Simulation

INTERVENTIONS:
Behavioral: Simulation — A 9-minute scenario based on an ACLS bradycardia algorithm in which a high-fidelity mannequin requires external pacing

SUMMARY:
The aim of this observational study is to compare the visual interests between residents in high-fidelity simulation practice

DETAILED DESCRIPTION:
Eighteen first year residents were asked to take part in a nine-minute scenario based on an ACLS bradycardia algorithm in which a high-fidelity mannequin required external pacing. The scenario was considered a success if the material was correctly set by the participant to obtain electrical and mechanical pacing in nine minutes. All participants were wearing Tobii Glasses® which is a mobile eye-tracking system that automatically aggregates gaze data. Infrared markers were placed in the simulation room to create Area of Interest (AOI), from which results were obtained. Three AOI were created: the vital signs monitor, the defibrillator/pacing unit and the head of the patient. Eye-tracking data were analyzed using the Tobii Studio® program.

ELIGIBILITY:
Inclusion Criteria:

* First-year residents from various specialties in their first three weeks of training

Exclusion Criteria:

* Underwent a previous residency
* Attending physicians in another country

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: First-year medical residents from various specialties at Université de Montréal Simulation center
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2016-07-18 (Actual); Study Completion 2017-01-25 (Actual)

PRIMARY OUTCOMES:
Time to first fixation, Total visit time | During the scenario
  Using eye-tracking technology, gaze date can be aggregate onto Areas of interest where data can be extrapolated.

CONTACTS AND LOCATIONS:
Overall Officials: Issam Tanoubi, Dr, Study Director — Université de Montreal; Mathieu Tourangeau, Dr, Principal Investigator — Université de Montreal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duchowski AT. A breadth-first survey of eye-tracking applications. Behav Res Methods Instrum Comput. 2002 Nov;34(4):455-70. doi: 10.3758/bf03195475. PMID 12564550
- [Background] Turgeon DP, Lam EW. Influence of Experience and Training on Dental Students' Examination Performance Regarding Panoramic Images. J Dent Educ. 2016 Feb;80(2):156-64. PMID 26834133
- [Background] Wilson MR, McGrath JS, Vine SJ, Brewer J, Defriend D, Masters RS. Perceptual impairment and psychomotor control in virtual laparoscopic surgery. Surg Endosc. 2011 Jul;25(7):2268-74. doi: 10.1007/s00464-010-1546-4. Epub 2011 Feb 27. PMID 21359902
- [Background] Schulz CM, Schneider E, Fritz L, Vockeroth J, Hapfelmeier A, Wasmaier M, Kochs EF, Schneider G. Eye tracking for assessment of workload: a pilot study in an anaesthesia simulator environment. Br J Anaesth. 2011 Jan;106(1):44-50. doi: 10.1093/bja/aeq307. Epub 2010 Oct 30. PMID 21037266
- [Background] Browning M, Cooper S, Cant R, Sparkes L, Bogossian F, Williams B, O'Meara P, Ross L, Munro G, Black B. The use and limits of eye-tracking in high-fidelity clinical scenarios: A pilot study. Int Emerg Nurs. 2016 Mar;25:43-7. doi: 10.1016/j.ienj.2015.08.002. Epub 2015 Oct 9. PMID 26455897